CLINICAL TRIAL: NCT01839240
Title: Phase I Investigation of the Feasibility of Combining 5-azacytidine With Highdose Cytarabine (HiDAC) and Mitoxantrone Chemotherapy in a Sequential Manner for Remission Induction in High-risk Acute Myelogenous Leukemia (AML)
Brief Title: Azacitidine, Cytarabine, and Mitoxantrone Hydrochloride in Treating Patients With High-Risk Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-0111; NCI-2012-02028 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-04-19; First posted 2013-04-24 (Estimated); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Azacitidine; Cytarabine; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (azacitidine, cytarabine, and mitoxantrone) (Experimental): INDUCTION: Patients receive azacitidine IV over 10-40 minutes or SC QD on days 1-5, cytarabine IV over 4 hours on days 6 and 10, and mitoxantrone hydrochloride IV over 60 minutes on days 6 and 10.
  CONSOLIDATION: Patients receive azacitidine IV over 10-40 minutes or SC QD on days 1-5. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients ineligible for allogeneic stem cell transplantation continue on to maintenance.
  MAINTENANCE: Patients receive azacitidine IV over 10-40 minutes or SC QD on days 1-5. Courses repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: azacitidine; Drug: cytarabine; Drug: mitoxantrone hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: azacitidine — Given IV or SC
  Other Names: 5-AC; 5-azacytidine; azacytidine; Vidaza
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: mitoxantrone hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Novantrone
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of azacitidine when given together with cytarabine and mitoxantrone hydrochloride in treating patients with high-risk acute myeloid leukemia. Drugs used in chemotherapy, such as azacitidine, cytarabine, and mitoxantrone hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Azacitidine may also help cytarabine and mitoxantrone hydrochloride work better by making the cancer cells more sensitive to the drugs

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the recommended phase II dose of 5-azacytidine (azacitidine) when combined with high-dose cytarabine (HiDAC) and mitoxantrone (mitoxantrone hydrochloride) chemotherapy in high-risk acute myeloid leukemia (AML) patients.

SECONDARY OBJECTIVES:

I. To determine the complete remission (CR) rate following the use of induction chemotherapy regimen of 5-azacytidine followed by high-dose cytarabine (HiDAC) and mitoxantrone chemotherapy in high-risk AML patients.

II. To determine the toxicity of the combination regimen. III. To determine the disease-free survival (DFS) and overall survival (OS) of the patient population.

IV. To determine the gene expression levels of topoisomerase II and deoxycytidine kinase in leukemia blasts pre-treatment and following therapy with 5-azacytidine.

V. To collect specimens for banking for use in future research studies with a view to elucidating the predictors of response to epigenetic therapies.

OUTLINE: This is a dose-escalation study of azacitidine.

INDUCTION: Patients receive azacitidine intravenously (IV) over 10-40 minutes or subcutaneously (SC) once daily (QD) on days 1-5, cytarabine IV over 4 hours on days 6 and 10, and mitoxantrone hydrochloride IV over 60 minutes on days 6 and 10.

CONSOLIDATION: Patients receive azacitidine IV over 10-40 minutes or SC QD on days 1-5. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients ineligible for allogeneic stem cell transplantation continue on to maintenance.

MAINTENANCE: Patients receive azacitidine IV over 10-40 minutes or SC QD on days 1-5. Courses repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following disease characteristics:

  * Therapy-related myeloid neoplasm (t-MN) age >= 18 years

    * Patients must have received cytotoxic chemotherapy, radiation, or a drug known to affect the properties of deoxyribonucleic acid (DNA) or cell growth, prior to current diagnosis of therapy-related myeloid neoplasm (t-MN); this broad definition is meant to include any prior therapy with chemicals that affect DNA replication, DNA integrity, or DNA structure, or chemicals that alter cell growth; this includes traditional cytotoxic chemotherapy, newer immunologic agents that have been shown to have cytotoxic activities in addition to immunosuppressive functions, and other chemicals; note that patients with primary AML could be diagnosed with a t- MN if morphology/cytogenetic analysis clearly indicated that the second process is not a relapse of the original disease
  * AML arising from an antecedent hematological disorder age >= 18 years
  * De novo AML in patients age >= 60 years
  * Relapsed and/or refractory AML >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment
* Male and female patients must use an effective contraceptive method during the study and for at least 6 months after study treatment
* Patients must be at least 2 weeks from major surgery, radiation therapy, participation in other investigational trials and must have recovered from clinically significant toxicities of these prior treatments
* Ability to understand and willingness to sign the informed consent form

Exclusion Criteria:

* Concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in this protocol
* Diagnosis of acute promyelocytic leukemia (APL)
* Use of investigational agents/any anticancer therapy within 2 weeks before study entry with the exception of hydroxyurea (note: for patients with hyperleukocytosis [white blood cell (WBC) > 20,000/uL], hydroxyurea [and leukapheresis, if clinically indicated] will be initiated and these patients will receive 5-azacytidine when the WBC count has decreased to =< 20,000/uL; hydroxyurea can be overlapped with 5-azacytidine in selected cases, after consultation with the study chair; hydroxyurea must be discontinued before the initiation of the HiDAC/mitoxantrone chemotherapy)
* Prior treatment with 5-azacytidine followed immediately by HiDAC and mitoxantrone as proposed in this study (note: prior therapy with 5-azacytidine or decitabine or HiDAC or mitoxantrone would be allowed-in patients with relapsed/refractory disease- unless the prior therapy was identical to the schema/schedule proposed in this study)
* Active second cancer other than specified; active cancer refers to cancer that requires systemic chemotherapy or biological therapy within 6 months of the study entry; patients who have received only hormonal therapy in the neoadjuvant or adjuvant setting in the past 6 months may participate in this study
* Have any other severe concurrent disease, or have a history of serious organ dysfunction (e.g. uncontrolled or severe cardiovascular disease, diabetes, pulmonary disease, infection, psychiatric illness) that may in the judgment of the treating physician/ principal investigator place the patient at undue risk to undergo treatment
* Pregnant or lactating patients
* Any significant concurrent illness that would, in the judgment of the treating physician/principal investigator, compromise patient safety or compliance, or study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06-06 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose of azacitidine when combined with high-dose cytarabine and mitoxantrone hydrochloride, based on incidence of dose limiting toxicity (DLT) graded according to the National Cancer Institute Common Toxicity Criteria, version 4 | 56 days
  DLT defined as any grade 4 or greater non-hematologic toxicity (except transient [less than 48 hours] nausea/vomiting, transient [less than 48 hours] liver function test derangements) or a grade 3 non-hematological toxicity lasting more than 7 days. Persistent bone marrow aplasia (in the absence of bone marrow involvement with disease) lasting more than 56 days would also be regarded as a DLT.

SECONDARY OUTCOMES:
Change in gene expression levels of topoisomerase II and deoxycytidine kinase in leukemic blasts pre-treatment and following therapy with azacitidine will be measured by real-time polymerase chain reaction (RT-PCR) | From baseline to day 56
  Will be compared using a two-sample t test. If the data do not appear to be normally distributed, a Wilcoxon rank sum test will be used in place of the t-test. Normality will be assessed using graphical techniques, such as normality probability plots.

CONTACTS AND LOCATIONS:
Overall Officials: Olatoyosi Odenike, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Cahill KE, Karimi YH, Karrison TG, Jain N, Green M, Weiner H, Fulton N, Kadri S, Godley LA, Artz AS, Liu H, Thirman MJ, Le Beau MM, McNerney ME, Segal J, Larson RA, Stock W, Odenike O. A phase 1 study of azacitidine with high-dose cytarabine and mitoxantrone in high-risk acute myeloid leukemia. Blood Adv. 2020 Feb 25;4(4):599-606. doi: 10.1182/bloodadvances.2019000795. PMID 32074275